CLINICAL TRIAL: NCT06157164
Title: Simultaneous UroLift™ and Holmium Laser Enucleation of the Prostatic Median Lobe for the Treatment of Benign Prostatic Hyperplasia in Men With Prominent Median Lobe Desiring Preservation of Ejaculation
Brief Title: IIT-2022-Simultaneous Urolift™ and Median Lobe Enucleation
Status: Terminated | Type: Observational
Why Stopped: Slow accrual
Sponsor: University of Kansas Medical Center (Other)
Responsible Party: Principal Investigator, Don Neff, MD, FACS, Principle Investigator, University of Kansas Medical Center
Other Study IDs: HSC 149327
Record Dates: First submitted 2023-09-28; First posted 2023-12-05 (Actual); Last update posted 2025-04-04 (Actual); Status verified 2025-04

CONDITIONS: Benign Prostatic Hyperplasia
Keywords: BPH
MeSH Terms: conditions — Prostatic Hyperplasia

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Simultaneous UroLift™ and HoLEP: UroLift System
  Interventions: Other: UroLift™ System and Holmium Laser Enucleation of the Prostate (HoLEP)

INTERVENTIONS:
Other: UroLift™ System and Holmium Laser Enucleation of the Prostate (HoLEP) — Simultaneous UroLift™ and Holmium Laser Enucleation of the Prostate (HoLEP) for the Treatment of BPH in Men with Prominent Median Lobe Desiring Preservation of Ejaculation

SUMMARY:
To evaluate postoperative outcomes of BPH/Lower urinary tract symptoms, erectile function, and ejaculatory capacity of simultaneous UroLiftTM and Holmium laser enucleation of the prostatic median lobe.

DETAILED DESCRIPTION:
Preserving ejaculation is a significant factor that impacts patient's decisions regarding what proceeding with treatment of BPH symptoms. The UroLiftTM system provides a safe procedure that has proven preservation of ejaculatory function. However, it is contraindicated in patients with prominent median lobes. The combination with laser median lobe enucleation may provide the same improvement in symptoms and widen patient inclusion criteria to those desire preserved ejaculation that also have a prominent median lobe.

ELIGIBILITY:
Inclusion Criteria:

1. Patients must be 45 years of age or older
2. Patients must be diagnosed with benign prostatic hyperplasia
3. Patients must opt for surgical management of their BPH with desire for preservation of ejaculatory function
4. Prominent median lobe with at least grade I intravesical protrusion of median lobe visualized on pre-operative cystoscopy

Exclusion Criteria:

1. Patients with baseline erectile and ejaculatory dysfunction as determined by a baseline IIEF-5 score < 15
2. Patients with a concomitant neurogenic bladder diagnosis (SCI, Parkinson, MS, cerebral palsy)
3. Patients with prostate glands greater or equal to 100 grams
4. Patients with less than a grade I intravesical protrusion of median lobe on pre-operative cystoscopy
5. Patients who are enrolled in other surgical or interventional trials at the time of this study are not eligible.

Min Age: 45 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Males 45 years of age or older who opt for surgical management of their BPH with desire for preservation of ejaculatory function.
Sampling Method: Non-Probability Sample
Enrollment: 3 (Actual)
Dates: Start 2023-02-06 (Actual); Primary Completion 2025-01-14 (Actual); Study Completion 2025-01-14 (Actual)

PRIMARY OUTCOMES:
International Prostate Symptom Score (IPSS) change (improvement) from baseline at 3 and 12 months. | Up to 12 months
  To evaluate improvement of symptoms through the International Prostate Symptom Score (IPSS) change (improvement) from baseline at 3 and 12 months.
  The IPSS is an 8-question screening tool used to screen for, rapidly diagnose, track the symptoms of, and suggest management of the symptoms of the disease benign prostatic hyperplasia (BPH).
  Scoring:
  0-7 Mildly symptomatic 8-19 Moderately symptomatic 20-35 Severely symptomatic

SECONDARY OUTCOMES:
Post-operative participant reported outcomes using benign prostatic hyperplasia impact index (BPHII). | Up to 12 months
  Evaluate post-operative participant reported outcomes using Benign Prostatic Hyperplasia Impact Index (BPHII). Post operative data will be compared to those values previously published for UroLift alone to evaluate non inferiority.
Post-operative participant reported outcomes using International Index of Erectile Function (IIEF). | Up to 12 months
  Evaluate post-operative sexual function using participant reported outcome International Index of Erectile Function (IIEF). Post operative data will be compared to those values previously published for UroLift alone to evaluate non inferiority.
Post-operative participant reported outcomes using Male Sexual Health Questionnaire for Ejaculatory Dysfunction Short Form (MSHQ-EjD-SF). | Up to 12 months
  Evaluate post-operative sexual function using participant reported outcome Male Sexual Health Questionnaire for Ejaculatory Dysfunction Short Form (MSHQ-EjD-SF). Post operative data will be compared to those values previously published for UroLift alone to evaluate non inferiority.
Post-Operative measurement of Peak Urine Flow Rate (Qmax) | Up to 12 months
  Evaluate post-operative lower urinary tract symptoms further with Peak Urine Flow Rate (Qmax). Post operative data will be compared to those values previously published for UroLift alone to evaluate non inferiority.
Post-Operative measurement of Post Void Residual (PVR) | Up to 12 months
  Evaluate post-operative lower urinary tract symptoms further with Post Void Residual (PVR). Post operative data will be compared to those values previously published for UroLift alone to evaluate non inferiority.

CONTACTS AND LOCATIONS:
Overall Officials: Donald Neff, Principal Investigator — University of Kansas Medical Center
Locations (1):
- University of Kansas Medical Center, Kansas City, Kansas, United States

IPD SHARING:
Plan to Share IPD: No